CLINICAL TRIAL: NCT01753713
Title: Phase II Study of TKI258 (Dovitinib) in Patients With Recurrent or Progressive Glioblastoma Who Have Progressed With or Without Anti-Angiogenic Therapy (Including Anti-VEGF Therapy)
Brief Title: Dovitinib in Treating Patients With Recurrent or Progressive Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Manmeet Ahluwalia, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Novartis (Industry)
Responsible Party: Sponsor-Investigator, Manmeet Ahluwalia, MD, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE4312; NCI-2012-02284 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-12-18; First posted 2012-12-20 (Estimated); Results first posted 2017-08-08 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-10

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one; Receptor Protein-Tyrosine Kinases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Anti-angiogenic Therapy Naive Patients (Experimental): Patients who have progressed without anti-angiogenic therapy. Patients receive dovitinib orally (PO) 5 days a week. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: dovitinib; Other: laboratory biomarker analysis
- Anti-angiogenic Therapy Patients (Experimental): Patients who have progressed on anti-angiogenic therapy. Patients receive dovitinib orally (PO) 5 days a week. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: dovitinib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: dovitinib — Given PO
  Other Names: CHIR-258; receptor tyrosine kinase (RTK) inhibitor TKI258; RTK inhibitor TKI258; TKI258
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well dovitinib works in treating patients with recurrent or progressive glioblastoma. Dovitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Anti-angiogenic Therapy Naive Patients: To determine 6 month progression-free survival (PFS6) in anti-angiogenic therapy (including anti-vascular endothelial growth factor (VEGF) therapy or bevacizumab) naive patients with recurrent glioblastoma (GBM) in patients treated with dovitinib

Anti-angiogenic Therapy Patients: To estimate time to progression in patients with recurrent or progressive Glioblastoma who have progressed on anti-angiogenic therapy (including anti-VEGF therapy).

SECONDARY OBJECTIVES:

1. To evaluate the side effect profile of dovitinib in both patient populations.
2. To evaluate the efficacy of dovitinib as measured by objective response rate (ORR) in both patient populations.
3. To estimate time to percentage of patients free from progression at 6 months (PFS-6)in patients with recurrent or progressive Glioblastoma who have progressed on antiangiogenic therapy (including anti-VEGF therapy). (Anti-angiogenic Therapy Patients)
4. To estimate time to progression in anti-angiogenic therapy (including anti-VEGF therapy or bevacizumab) naiVe patients with recurrent glioblastoma (GBM) in patients treated with dovitinib. (Anti-angiogenic Therapy Naive Patients)
5. To evaluate the overall survival (OS) in both patient populations.

EXPLORATORY OBJECTIVES:

To explore association between clinical outcome and potential biomarkers that may include microparticles, PlGF, PDGF-AA, PDGF-AB, PDGF-BB, SDF-1a, thrombospondin-1, Ang1, and Il-6, IL-8 and FGF.

OUTLINE:

Patients receive dovitinib orally (PO) 5 days a week. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed glioblastoma, recurrent after standard external-beam fractionated radiotherapy and temozolomide chemotherapy
* Patients who have NOT received any anti-angiogenic therapy (Anti-VEGF, including avastin, cediranib, or other anti-angiogenic therapies like cilengitide) on Anti-angiogenic Therapy Naive Patients Arm. No more than two recurrences are allowed on Anti-angiogenic Therapy Naive Patients Arm.
* Patients who have received any anti-angiogenic therapy (Anti-VEGF, including avastin, cediranib, or other anti-angiogenic therapies like cilengitide) on Anti-angiogenic Therapy Patients Arm. Any number of recurrences are allowed on Anti-angiogenic Therapy Patients Arm.
* Karnofsky performance status ≥ 60%
* Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
* Platelets ≥ 100 x 10^9/L
* Hemoglobin (Hgb) > 9 g/dL
* Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0 x ULN
* Serum creatinine ≤ 1.5 x ULN
* Minimum interval since completion of radiation treatment is 12 weeks
* Minimum interval since last drug therapy 2 weeks since last non-cytotoxic therapy 3 weeks must have elapsed since the completion of a non-nitrosourea containing chemotherapy regimen 6 weeks since the completion of a nitrosourea containing chemotherapy regimen
* Patients must be able to provide written informed consent
* Patients with the potential for pregnancy or impregnating their partner must agree to follow acceptable birth control methods to avoid conception; the anti-proliferative activity of this experimental drug may be harmful to the developing fetus or nursing infant; female patients of child-bearing potential must have a negative pregnancy test
* Patients must have no concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix and breast, adequately treated stage I or II cancer from which the patient is in complete remission; patients with other prior malignancies must be disease-free for ≥ three years
* Patients must be maintained on a stable corticosteroid regimen from the time of their baseline scan until the start of treatment and/or for at least 5 days before starting treatment

Exclusion Criteria:

* Patients who have undergone major surgery (e.g. intra-thoracic, intra-abdominal or intra-pelvic), open biopsy or significant traumatic injury ≤ 4 weeks prior to starting study drug, or patients who have had minor procedures, percutaneous biopsies or placement of vascular access device ≤ 1 week prior to starting study drug, or who have not recovered from side effects of such procedure or injury
* Patients with a history of pulmonary embolism (PE), or untreated deep venous thrombosis (DVT) within the past 6 months
* Patients with any of the following concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study:

  * Impaired cardiac function or clinically significant cardiac diseases, including any of the following:

    * History or presence of serious uncontrolled ventricular arrhythmias
    * Clinically significant resting bradycardia
    * Left ventricular ejection fraction (LVEF) assessed by 2-dimensional (2-D) echocardiogram (ECHO) < 50% or lower limit of normal (whichever is higher) or multi gated acquisition scan (MUGA) < 45% or lower limit of normal (whichever is higher)
    * Any of the following within 6 months prior to starting study drug: myocardial infarction (MI), severe/unstable angina, coronary artery bypass graft (CABG), congestive heart failure (CHF), cerebrovascular accident (CVA), and transient ischemic attack (TIA)
    * Uncontrolled hypertension defined by a systolic blood pressure (SBP) ≥ 160 mm Hg and/or diastolic blood pressure (DBP) ≥ 100 mm Hg, with or without anti-hypertensive medication(s)
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of dovitinib (e.g. ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* Cirrhosis, chronic active hepatitis or chronic persistent hepatitis
* Known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory)
* Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g. active or uncontrolled infection, uncontrolled diabetes) that could cause unacceptable safety risks or compromise compliance with the protocol
* Women of child-bearing potential, who are biologically able to conceive, not employing two forms of highly effective contraception; highly effective contraception (e.g. male condom with spermicide, diaphragm with spermicide, intra-uterine device) must be used by both sexes during the study and must be continued for 8 weeks after the end of study treatment; oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study; women of child-bearing potential, defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (e.g., who has had menses any time in the preceding 12 consecutive months), must have a negative serum pregnancy test ≤ 14 days prior to starting study treatment
* Fertile males not willing to use contraception, as stated above
* Patients who are currently receiving full dose anticoagulation treatment with therapeutic doses of warfarin or anti-platelet therapy (e.g., Plavix [clopidogrel bisulfate]); treatment with locally accepted low molecular weight heparin and low dose of acetylsalicylic acid (i.e., 81mg or 100 mg daily) to prevent cardiovascular events or strokes is allowed
* Patients unwilling or unable to comply with the protocol
* Any significant hemorrhage defined as > 1 cm diameter of blood seen on the MRI or CT scan. If > 1 cm of acute blood is detected, the patient will be ineligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-12-20 (Actual); Primary Completion 2015-01-28 (Actual); Study Completion 2017-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manmeet Ahluwalia, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anti-angiogenic Therapy Patients | Anti-angiogenic Therapy Naive Patients
Started | 14 | 19
Completed | 14 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anti-angiogenic Therapy Naive Patients | Anti-angiogenic Therapy Patients | Total
Number analyzed (Participants) | 19 | 14 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 13 | 29
  >=65 years | 3 | 1 | 4
Age, Continuous [Median (Full Range); unit: years] | 58 [33 to 68] | 51 [26 to 66] | 57 [26 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 12 | 9 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 13 | 32
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 1 | 2
  White | 16 | 11 | 27
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 14 | 33

OUTCOME MEASURES:

1. Primary Outcome: Arm 1: Progression Free Survival (PFS)
Description: Number of anti-angiogenic therapy (including anti-VEGF therapy or bevacizumab) naive patients with recurrent glioblastoma (GBM). The progression- free survival (PFS) at 6 months is defined as the time from randomization to objective tumor progression or death. So patients who have CR, PR or SD at 6 months will constitute PFS-6. Progression is defined using the Response Assessment in Neuro-Oncology (RANO) Criteria where CR = Total disappearance of lesions, PR = >50% reduction in lesions and SD = <25% reduction in lesions
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-angiogenic Therapy Naive Patients | Anti-angiogenic Therapy Patients
Number analyzed (Participants) | 19 | 14
Participants | 0 | 0

2. Primary Outcome: Arm 2: Determine Median Time to Progression
Description: Anti-angiogenic therapy (including anti-VEGF therapy or bevacizumab) patients with recurrent glioblastoma (GBM). Time to tumor progression (TTP), is defined as the time from randomization to time of progressive disease. So it is ongoing and will be assessed every 8 weeks …8, 16, 24, 32 …week. Progression is defined as >25% increase in size of lesions or evidence of new lesions
Time Frame: From randomization to time of progression every 8 weeks (2 cycles of treatment) up to 32 weeks
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Anti-angiogenic Therapy Naive Patients | Anti-angiogenic Therapy Patients
Number analyzed (Participants) | 19 | 14
Months | 1.8 [1.3 to 2.8] | 1.8 [0.7 to 1.8]

3. Secondary Outcome: Toxicity Assessed Using Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Description: Number of adverse events in patients in both populations (grade 1-5). Grade 1 are defined as mild events characterized as asymptomatic or mild symptoms; clinical or diagnostic observations only; no intervention indicated. Grade 2 are moderate events with minimal, local or non invasive interventions indicated. Grade 3 are severe or medically significant events but not immediately life-threatening; hospitalization indicated. Grade 4 are life-threatening consequences with urgent intervention indicated. Grade 5 are deaths related to events
Time Frame: Assessed until 30 days after treatment up to 32 weeks
Measure: Number; unit: Events
Arm/Group | Anti-angiogenic Therapy Naive Patients | Anti-angiogenic Therapy Patients
Number analyzed (Participants) | 19 | 14
Events
  Grade 1 | 217 | 119
  Grade 2 | 109 | 85
  Grade 3 | 55 | 40
  Grade 4 | 2 | 5
  Grade 5 | 1 | 2

4. Secondary Outcome: Objective Response Rate Using Modified Revised Assessment in Neuro-Oncology (RANO) Criteria
Description: Number of patients (both populations) with a complete response (CR-no measurable disease), partial response (PR >50% reduction in measurable disease), minor response (MR >25% reduction of measurable disease), stable disease (SD <25% reduction) and progressive disease (PD >25% measurable disease and new lesions).
Time Frame: Up to 30 days after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-angiogenic Therapy Naive Patients | Anti-angiogenic Therapy Patients
Number analyzed (Participants) | 19 | 14
Participants
  Complete Response | 0 | 0
  Progressive Disease | 8 | 8
  Stable Disease | 3 | 2
  Unknown | 6 | 4
  Partial Response | 2 | 0

5. Secondary Outcome: Median Progression Free Survival
Description: The progression- free survival (PFS) at 6 months is defined as the time from randomization to objective tumor progression or death. So patients who have CR, PR or SD at 6 months will constitute PFS-6
Time Frame: 6 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Anti-angiogenic Therapy Naive Patients | Anti-angiogenic Therapy Patients
Number analyzed (Participants) | 19 | 14
Months | 2.0 [1.3 to 3.7] | 1.8 [0.9 to 1.8]

6. Secondary Outcome: Overall Survival
Description: The Kaplan-Meier method will be used. Overall survival is defined as the time from randomization to death.
Time Frame: to death, approximately 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Anti-angiogenic Therapy Naive Patients | Anti-angiogenic Therapy Patients
Number analyzed (Participants) | 19 | 14
Months | 8.0 [4.4 to 11.7] | 4.3 [2.6 to 6.7]

7. Other Pre Specified Outcome: Changes From Baseline in Circulating Growth Factors and Soluble Receptors.
Description: To assess the pharmacodynamic effect of dovitinib on potential plasma biomarkers that may include measuring concentrations of circulating, microparticles, PlGF, PDGF-AA, PDGF-AB, PDGF-BB, SDF-la, thrombospondin-l, Angl, and 11-6, IL-8 and FGF.
Time Frame: Up to 30 days after treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: adverse events were monitored for at least 30 days following the last dose of treatment. For this study, the maximum time following a subject was 2 years.
Arm/Group | Anti-angiogenic Therapy Naive Patients | Anti-angiogenic Therapy Patients
All-Cause Mortality (participants affected / at risk) | 1/19 | 2/14
Serious Adverse Events (participants affected / at risk) | 10/19 | 7/14
Other Adverse Events (participants affected / at risk) | 19/19 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-angiogenic Therapy Naive Patients (N=19) | Anti-angiogenic Therapy Patients (N=14)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death NOS (General disorders) | 1 (1) | 2 (2)
Fever (General disorders) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 2 (3) | 1 (1)
Confusion (Psychiatric disorders) | 3 (4) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 6 (6) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-angiogenic Therapy Naive Patients (N=19) | Anti-angiogenic Therapy Patients (N=14)
Alanine aminotransferase increased (Investigations) | 12 (16) | 11 (15)
Platelet count decreased (Investigations) | 13 (17) | 10 (19)
Lymphocyte count decreased (Investigations) | 12 (20) | 6 (8)
Aspartate aminotransferase increased (Investigations) | 5 (9) | 6 (8)
Lipase increased (Investigations) | 7 (12) | 4 (6)
Cholesterol high (Investigations) | 6 (6) | 4 (4)
White blood cell decreased (Investigations) | 6 (7) | 4 (5)
Serum amylase increased (Investigations) | 5 (5) | 2 (3)
Weight loss (Investigations) | 1 (1) | 4 (4)
Neutrophil count decreased (Investigations) | 2 (4) | 2 (3)
GGT increased (Investigations) | 0 (0) | 2 (2)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Weight gain (Investigations) | 1 (1) | 0 (0)
Fatigue (General disorders) | 12 (28) | 7 (10)
Gait disturbance (General disorders) | 5 (8) | 3 (4)
Edema limbs (General disorders) | 3 (4) | 1 (2)
Fever (General disorders) | 4 (9) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0)
Edema face (General disorders) | 1 (1) | 1 (2)
Localized edema (General disorders) | 2 (2) | 0 (0)
Facial pain (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (3) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 15 (21) | 9 (15)
Hypokalemia (Metabolism and nutrition disorders) | 4 (5) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 9 (15) | 9 (10)
Nausea (Gastrointestinal disorders) | 10 (15) | 2 (3)
Vomiting (Gastrointestinal disorders) | 4 (6) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 4 (5)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (3) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 10 (17) | 3 (5)
Dysphasia (Nervous system disorders) | 3 (3) | 2 (3)
Seizure (Nervous system disorders) | 4 (7) | 1 (3)
Dysgeusia (Nervous system disorders) | 3 (4) | 1 (1)
Dysarthria (Nervous system disorders) | 2 (2) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 2 (2)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Concentration impairment (Nervous system disorders) | 0 (0) | 1 (1)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (11) | 4 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 4 (8) | 4 (8)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (5) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 7 (10) | 2 (3)
Hypertension (Vascular disorders) | 1 (1) | 5 (9)
Proteinuria (Renal and urinary disorders) | 3 (3) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 3 (4)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (2) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (5) | 1 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (6) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (3) | 2 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 4 (5) | 2 (3)
Bruising (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes